CLINICAL TRIAL: NCT07046884
Title: Improving Personalized Treatment in Oncology: Effects of Integrated Oncological Decision-making
Acronym: IPTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, lwelling, Dr. L. Welling, Leiden University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N23.071
Record Dates: First submitted 2024-09-30; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Oncology
Keywords: Oncology; Integrated Care; Personalized treatment; Shared decision-making
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will use a stepped-wedge cluster randomized trial design. Eight oncological care paths (clusters) will transition from current practice (control) to a locally tailored IODM-based practice (intervention condition) in four steps (two clusters per step), where order is determined by randomization.
Who Masked: Participant
Masking Description: Participants will not know whether their onocolgical care pathway has already integrated the IODM (intervention) or is practising care as usual (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Current care pathway (Control condition) (No Intervention): In this arm the participants receive care as usual.
- IODM integrated care pathway (Active Comparator): In this arm the participants receive care within an oncological care path that has integrated the IODM within their daily practice
  Interventions: Behavioral: Integrated Oncological Decision-making Model

INTERVENTIONS:
Behavioral: Integrated Oncological Decision-making Model — In the IODM-based practice, the following three information components should be incorporated when forming a personalized treatment plan: 1. State-of-the-art oncological treatment options with advantages and disadvantages; 2. General health status based on physical, psychosocial, and emotional functioning; 3. Goals and preferences of the patient, both in treatment and daily life. Together with the professionals, optimal tools and strategies to integrate these components within the care path will be discussed.
  Arms: IODM integrated care pathway

SUMMARY:
The research aims to evaluate an Integrated Oncological Decision-making Model (IODM) to tailor oncological treatment plans to individual patients. The primary objective is to assess the impact of the IODM on personalized decision-making and patient outcomes. The study will employ a stepped-wedge cluster randomized trial design involving eight oncological care paths across four medical centers in the Netherlands. The study population consists of 400 adult patients (50 per care path) who will undergo treatment based on either standard clinical guidelines (control) or the IODM (intervention). The intervention involves integrating three key components: oncological treatment options, patient's general health status, and patient's goals and preferences. The main study parameters include measuring the discordance between recommendations based on medical information and final treatment decisions, assessing whether discordance reflects more personalized decision-making, and evaluating the implementation process of the IODM.

DETAILED DESCRIPTION:
Rationale: Currently, oncological treatment plans and decision-making are predominantly based on medical information following strict guidelines. Based on the conviction that oncological treatment plans can and should be more tailored to the individual, an outline for the Integrated Oncological Decision-making Model (IODM) has been developed. The IODM aims to individualize treatment decisions through the integration of patient's health status and goals/preferences in formulating treatment decisions.

Objectives: The primary objective of the current study is to evaluate the effect of the IODM on personalized decision-making and patient outcomes. We hypothesize that with the use of the IODM, decisions will more often differ from treatment recommendation based on clinical guidelines only, and that use of the IODM intervention will lead to more personalized decisions. The secondary objective of this study is to perform an extensive process evaluation of the implementation and strategies of the IODM.

Study design: The study will use a stepped-wedge cluster randomized trial design. Eight oncological care paths (clusters) will transition from current practice (control) to a locally tailored IODM-based practice (intervention condition) in four steps (two clusters per step), where order is determined by randomization.

Study population: Study participants will be a convenience sample of patients (n=400 total, n=50 per care path) from two oncological care paths per center, in four medical centers (LUMC, UMCG, MUMC+ and Zuyderland) in the Netherlands. The minimal age of participants is 18.

Intervention: In the IODM-based practice, the following three information components should be incorporated when forming a personalized treatment plan: 1. State-of-the-art oncological treatment options with advantages and disadvantages; 2. General health status based on physical, psychosocial, and emotional functioning; 3. Goals and preferences of the patient, both in treatment and daily life. Together with the professionals, optimal tools and strategies to integrate these components within the care path will be discussed.

Main study parameters/endpoints: Our primary outcome is the discordance between the treatment recommendation based on clinical guidelines and the final treatment decision. We will measure whether discordance is due to more personalized decision-making, using shared decision-making outcome measures, and assessment of IODM components.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age = 18+
* Patient is included in participating oncological care path
* Patient does not yet have a treatment plan
* Patient, partner, or caregiver who reads and speaks Dutch sufficiently to understand the research material and to complete the questionnaires
* Patient must be able to participate in the decision-making process

Exclusion Criteria:

• Patient, partner, or caregiver cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients with Discordance Between Standard Treatment Recommendation and Actual Treatment Decision | During the duration of the trial including 12-month follow-up (2 years)
  This outcome measures the proportion of patients for whom the actual treatment decision deviates from the standard treatment recommendation based solely on medical-technical information. The standard treatment recommendation is defined in advance by oncology teams using medical-technical criteria (e.g., tumor type, stage, comorbidities), and is either collected prospectively from multidisciplinary tumor boards or derived from guideline-based recommendations documented in the electronic health record (EHR). The actual treatment decision is the treatment option selected by the clinical team and/or patient during the decision-making process, regardless of whether this treatment is ultimately delivered. Discordance is defined as any difference between the standard treatment recommendation and the actual treatment decision. This outcome will be used to evaluate whether implementing the IODM intervention, designed to support more personalized care, is associated with a change in discordance

SECONDARY OUTCOMES:
Cancer-Related Quality of Life Assessed Using the EORTC QLQ-C30 Questionnaire | 2 years
  Quality of life is measured using the EORTC QLQ-C30 questionnaire, which evaluates multiple domains: physical, role, cognitive, emotional, and social functioning; symptom scales such as fatigue and pain; and global health status. Scores range from 0 to 100. Higher scores indicate better functioning or health on functional and global scales, and greater symptom severity on symptom scales.
Age of Participants at Time of Enrollment (Years) | 2 years
  Age is recorded in years based on participant self-report or medical records at the time of enrollment in the study. Data will be reported as mean, median, and range.
Frailty Assessed Using the Clinical Frailty Scale (CFS) | 2 years
  Frailty is measured using the Clinical Frailty Scale (CFS), a clinician-reported tool that assesses a patient's vulnerability to adverse health outcomes based on their physical and cognitive condition. The scale ranges from 1 to 9, where 1 indicates very fit and 9 indicates terminally ill. Higher scores reflect greater frailty.
Resilience Assessed Using the Brief Resilience Scale (BRS) | 2 years
  Resilience is measured using the Brief Resilience Scale (BRS), a patient-reported questionnaire designed to assess the ability to recover from stress. The scale ranges from 1 to 5, with higher scores indicating greater resilience.
Optimism Assessed Using the Life Orientation Test-Revised (LOT-R) | 2 years
  Optimism is measured using the Life Orientation Test-Revised (LOT-R), a patient-reported questionnaire that assesses an individual's general tendency toward optimism versus pessimism. Scores range from 0 to 24, with higher scores indicating greater optimism.
Mean Score on Quality of Life Impact of Symptoms Assessed with EORTC QLQ-C30 and Additional Items (coping with side effects) | 2 years
  This outcome measures how well patients cope with side effects from cancer treatment, operationalized as the self-reported impact of symptoms on various quality of life (QoL) domains. Symptoms are identified using disease-specific EORTC questionnaires. The impact of these symptoms is measured using items from the EORTC QLQ-C30 Core Quality of Life questionnaire, supplemented with additional questions covering domains not fully captured by the QLQ-C30, including physical functioning, emotional well-being, independence, social relationships, meaning in life, and daily activities. Scores are aggregated by calculating mean scores per domain and overall, with higher scores indicating greater impact and therefore lower coping effectiveness.
Shared Decision-Making Assessed Using the I-Share Questionnaire | 2 years
  Shared decision-making is measured using the 5-Likert scale, 17-item I-Share questionnaire, a patient-reported outcome measure that assesses the patient's experience of shared decision-making during medical consultations. Higher scores indicate a greater perceived level of shared decision-making.
Decisional Conflict Assessed Using the Decisional Conflict Scale | 2 years
  Decisional conflict is measured using the Decisional Conflict Scale, a patient-reported questionnaire that evaluates uncertainty and perceived difficulty in making a health-related decision. Scores range from 0 to 100, with higher scores indicating greater decisional conflict. 16 item 5 response categories.
Decision Regret Assessed Using the Decision Regret Scale | 2 years
  Decision regret is measured using the Decision Regret Scale, a patient-reported questionnaire that assesses the level of regret a patient feels after making a health-related decision. Scores range from 0 to 100, with higher scores indicating greater decision regret. 5 items, 5 answer categories
Patient Role Preference Assessed Using the Modified Control Preference Scale | 2 years
  The Modified Control Preference Scale is a patient-reported measure that assesses the patient's perceived and preferred role in the treatment decision-making process. Responses are categorized into three groups reflecting whether the patient prefers a passive role (decision made by the clinician), a shared role (decision made together with the clinician), or an active role (decision made primarily by the patient). 1-Item, 5 categories.
Type of Companion Present During Treatment Decision Consultation as Recorded in the Electronic Medical Record (EMR) | 2 years
  This outcome records the type of companion (e.g., partner, child, friend, or other caregiver) who was present during the treatment decision consultation. Information is extracted from the electronic medical record (EMR), where the presence and relationship of companions are noted by clinical staff when available. Data will be reported as counts per companion type.
Shared Decision-Making Assessed Using Observational Coding with the 4SDM Framework | 2 years
  Shared decision-making is measured through researcher-coded audio recordings of clinical consultations, using the 4SDM observational framework. The coding assesses the extent to which shared decision-making principles were applied during the consultation, including steps such as team talk, option talk, preference talk, and decision talk.
Patients' Perception of Patient-Centeredness Assessed Using a Patient-Reported Questionnaire | 2 years
  Patient-centeredness is measured using a patient-reported questionnaire that assesses the extent to which patients perceive their care as aligned with their individual values, needs, and preferences. Scores indicate the degree of patient-centeredness experienced, with higher scores reflecting a greater perception of personalized, respectful, and responsive care.
Participant Sex as Recorded in the Electronic Medical Record (EMR) | 2 years
  Sex is recorded as part of routine clinical documentation and extracted from the electronic medical record (EMR). Categories include: male and female. Data will be reported as the number of participants in each category.
Migration Background Based on Self-Reported Country of Birth and Parental Origin | 2 years
  Migration background is determined based on self-reported data on the participant's own country of birth and the countries of birth of both parents. Participants are categorized according to national guidelines into groups such as: no migration background, first-generation migrant (participant born abroad), or second-generation migrant (participant born in the reporting country with at least one parent born abroad). Data will be reported as counts per category.
ighest Level of Education Completed as Self-Reported by Participant | 2 years
  Education level is measured based on self-reported data from participants indicating the highest level of education they have completed. Categories include, for example: primary education, secondary education, vocational training, and higher education (e.g., university or equivalent). Data will be reported as the number of participants in each education category.
Living Situation as Self-Reported by Participant | 2 years
  Living situation is measured using self-reported data from participants, indicating with whom they live. Response categories include: living alone, living with a partner, living with family (e.g., children or parents), or living with others (e.g., housemates, caregivers). Data will be reported as the number of participants in each category.
Health Literacy Assessed Using a Three-Item Dutch Version of the SBS-Q | 2 years
  Health literacy is measured using a three-item Dutch version of the Set of Brief Screening Questions (SBS-Q), a patient-reported questionnaire that assesses an individual's ability to understand and use health-related information. Each item is scored on a 5-point Likert scale. Responses are combined into an overall score, with higher scores indicating lower health literacy. Data will be reported as mean scores and/or categorized into levels of health literacy (e.g., adequate vs. inadequate).
Activities of Daily Living using Katz ADL | 2 years
  Description: Functional independence in basic activities of daily living is assessed using the Katz ADL Index, a patient-reported measure. The Katz ADL evaluates the ability to perform tasks such as bathing, dressing, toileting, transferring, continence, and feeding.
  Scoring: The Katz ADL provides scores ranging from 0 (completely dependent) to 6 (completely independent), with higher scores indicating greater independence.
Type of Tumour Working Group Involved in the Case as Recorded in the Medical Record | 2 years
  This outcome captures which multidisciplinary tumour working group (e.g., breast, lung, gastrointestinal) was responsible for managing each case. The data are extracted from the medical record or tumour board documentation. Each participant is assigned to a tumour working group based on their primary diagnosis. Data will be reported as the number of participants per tumour group.
Histological or Pathological Tumor Type as Recorded in the Medical Record | 2 years
  The tumor type is classified based on histological or pathological examination results documented in the medical record. Tumors are categorized according to established classification systems relevant to the cancer type (e.g., adenocarcinoma, squamous cell carcinoma). Data will be reported as counts per tumor type category.
verall Tumor Stage Assessed Using the TNM Classification | 2 years
  The overall stage of the cancer is determined according to the TNM classification system, based on tumor size (T), lymph node involvement (N), and presence of metastases (M). Stages are categorized from I to IV, with higher stages indicating more advanced disease. Data will be reported as the number of participants in each stage category.
TNM Score Based on Tumor Size, Lymph Node Involvement, and Metastasis | 2 years
  The TNM score summarizes cancer staging by evaluating three components: T (tumor size and extent), N (lymph node involvement), and M (presence of distant metastases). Each component is assessed according to standard clinical criteria. The combined TNM score is used to classify disease severity and guide treatment decisions. Data will be reported as individual T, N, and M categories and as overall stage groups.
Name of Hospital Providing Patient Care as Recorded in the Electronic Medical Record (EMR) | 2 years
  The hospital where the patient receives care is recorded in the electronic medical record (EMR). This information provides context regarding the healthcare setting and available infrastructure. Data will be reported as counts of patients per hospital.
Number and Type of Clinicians Involved in Patient Care as Extracted from the Electronic Medical Record | 2 years
  The number and types of clinicians involved in each patient's care are extracted from the electronic medical record (EMR). This includes consultations and interactions with various specialists such as oncologists, surgeons, radiologists, palliative care specialists, and others. Data will be reported as the total number of clinicians seen per patient and as a breakdown by clinician specialty.
Primary Treatment Decision Consultation as Recorded in the Electronic Medical Record (EMR) | 2 years
  This outcome captures details of the specific clinical consultation during which the primary treatment decision was made, as documented in the EMR. Data include the date of the consultation and the context/type of decision discussed, such as surgery, chemotherapy, or palliative care. This identifies the critical discussion shaping the patient's care plan.
Primary Clinician Responsible for Patient Care as Recorded in the Electronic Medical Record (EMR) | 2 years
  The primary clinician responsible for managing the patient's care is identified based on documentation in the EMR. This includes the clinician's name, medical specialty (e.g., oncologist, surgeon), and their role in coordinating treatment and decision-making for the patient.

OTHER OUTCOMES:
Feasibility of Implementing the IODM Intervention Assessed by Healthcare Professional Questionnaire | 2 years
  Feasibility is assessed by evaluating how practical and easy it is to integrate the IODM intervention into routine oncological care workflows. Healthcare professionals complete a questionnaire measuring whether the intervention can be consistently and effectively used without disrupting existing processes. Data will be reported as summary scores from the questionnaire.
Appropriateness of the IODM Intervention as Assessed by Healthcare Professionals | 2 years
  Appropriateness measures the extent to which the IODM intervention aligns with clinical needs, goals of healthcare professionals, and existing oncological care pathway guidelines. It reflects how well the intervention fits within the clinical context. Data are collected via a questionnaire completed by healthcare professionals using a standardized assessment tool.
Acceptability of the Integrated Oncology Decision-Making Model (IODM) Assessed by Healthcare Professionals | 2 years
  Acceptability refers to the extent to which healthcare professionals perceive the IODM intervention as satisfactory and suitable for use in oncological care. This includes their overall perception of its value and usefulness in clinical practice. Data are collected via the Acceptability of Intervention Measure (AIM) questionnaire completed by healthcare professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Lieke Welling, MD PhD (Dr), Principal Investigator — Department of Surgery
Locations (4):
- Netherlands (4):
  - University Medical Center Groningen (UMCG), Groningen
  - Leiden University Medical Center (LUMC), Leiden
  - Maastricht University Medical Center, Maastricht
  - Zuyderland MC, Sittard

IPD SHARING:
Plan to Share IPD: No
Data will only be shared among researchers within the consortium

REFERENCES:
- [Background] Bomhof-Roordink H, Stiggelbout AM, Gartner FR, Portielje JEA, de Kroon CD, Peeters KCMJ, Neelis KJ, Dekker JWT, van der Weijden T, Pieterse AH; iSHARE Study group. Patient and physician shared decision-making behaviors in oncology: Evidence on adequate measurement properties of the iSHARE questionnaires. Patient Educ Couns. 2022 May;105(5):1089-1100. doi: 10.1016/j.pec.2021.08.034. Epub 2021 Aug 28. PMID 34556384
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. Fam Med. 2004 Sep;36(8):588-94. PMID 15343421
- [Background] Festen S, Kok M, Hopstaken JS, van der Wal-Huisman H, van der Leest A, Reyners AKL, de Bock GH, de Graeff P, van Leeuwen BL. How to incorporate geriatric assessment in clinical decision-making for older patients with cancer. An implementation study. J Geriatr Oncol. 2019 Nov;10(6):951-959. doi: 10.1016/j.jgo.2019.04.006. Epub 2019 Apr 26. PMID 31031193
- [Background] Festen S, van der Wal-Huisman H, van der Leest AHD, Reyners AKL, de Bock GH, de Graeff P, van Leeuwen BL. The effect of treatment modifications by an onco-geriatric MDT on one-year mortality, days spent at home and postoperative complications. J Geriatr Oncol. 2021 Jun;12(5):779-785. doi: 10.1016/j.jgo.2020.12.003. Epub 2020 Dec 17. PMID 33342722
- [Background] Hamaker ME, Te Molder M, Thielen N, van Munster BC, Schiphorst AH, van Huis LH. The effect of a geriatric evaluation on treatment decisions and outcome for older cancer patients - A systematic review. J Geriatr Oncol. 2018 Sep;9(5):430-440. doi: 10.1016/j.jgo.2018.03.014. Epub 2018 Apr 7. PMID 29631898
- [Background] Hansson E, Ekman I, Swedberg K, Wolf A, Dudas K, Ehlers L, Olsson LE. Person-centred care for patients with chronic heart failure - a cost-utility analysis. Eur J Cardiovasc Nurs. 2016 Jun;15(4):276-84. doi: 10.1177/1474515114567035. Epub 2015 Jan 16. PMID 25595358
- [Background] Stiggelbout AM, Pieterse AH, De Haes JC. Shared decision making: Concepts, evidence, and practice. Patient Educ Couns. 2015 Oct;98(10):1172-9. doi: 10.1016/j.pec.2015.06.022. Epub 2015 Jul 15. PMID 26215573
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Scheier MF, Carver CS. Optimism, coping, and health: assessment and implications of generalized outcome expectancies. Health Psychol. 1985;4(3):219-47. doi: 10.1037//0278-6133.4.3.219. PMID 4029106
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Reynolds A. Patient-centered Care. Radiol Technol. 2009 Nov-Dec;81(2):133-47. PMID 19901351
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Maizes V, Rakel D, Niemiec C. Integrative medicine and patient-centered care. Explore (NY). 2009 Sep-Oct;5(5):277-89. doi: 10.1016/j.explore.2009.06.008. PMID 19733814
- [Background] Lamb BW, Brown KF, Nagpal K, Vincent C, Green JS, Sevdalis N. Quality of care management decisions by multidisciplinary cancer teams: a systematic review. Ann Surg Oncol. 2011 Aug;18(8):2116-25. doi: 10.1245/s10434-011-1675-6. Epub 2011 Mar 26. PMID 21442345
- [Background] Kaasa S, Bjordal K, Aaronson N, Moum T, Wist E, Hagen S, Kvikstad A. The EORTC core quality of life questionnaire (QLQ-C30): validity and reliability when analysed with patients treated with palliative radiotherapy. Eur J Cancer. 1995 Dec;31A(13-14):2260-3. doi: 10.1016/0959-8049(95)00296-0. PMID 8652253
- [Background] Janz NK, Wren PA, Copeland LA, Lowery JC, Goldfarb SL, Wilkins EG. Patient-physician concordance: preferences, perceptions, and factors influencing the breast cancer surgical decision. J Clin Oncol. 2004 Aug 1;22(15):3091-8. doi: 10.1200/JCO.2004.09.069. PMID 15284259
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207